CLINICAL TRIAL: NCT06067581
Title: Clinical Study on the Safety and Efficacy of SENL103 Autologous T Cell Injection in the Treatment of Recurrent or Refractory Plasma Cell Blood Tumors
Brief Title: the Safety and Efficacy of SENL103 Autologous T Cell Injection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENL103 CAR-T
Record Dates: First submitted 2023-08-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: BCMA
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART (Experimental): This study will follow the classic "3+3" design and increase the dose according to three dose groups. Each dose group will have 3-6 eligible subjects selected according to the inclusion/exclusion criteria, with a dose of 1.0 × 10^6, 2.0 × 10^6, 3.0 × Increase the dose by 10^6 CAR-T cells/kg.
  Interventions: Biological: SENL103

INTERVENTIONS:
Biological: SENL103 — Patients will be treated with BCMA CAR-T cells

SUMMARY:
To observe the safety and efficacy of SENL103 cells in the treatment of patients with recurrent or refractory plasma cell blood tumors.

DETAILED DESCRIPTION:
Primary endpoint To observe the number and incidence of adverse events after intravenous infusion of SENL103. To evaluate possible adverse reactions recorded within 1 month after SENL103 infusion, including the number, incidence and severity of symptoms such as cytokine release syndrome and neurotoxic reactions; Secondary endpoints

1. Efficacy indicators: The efficacy after cell retransfusion was observed by strict complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), stable disease (SD), and progression-free survival (PFS rate);
2. PK index: the highest concentration of SENL103 cells amplified in peripheral blood (Cmax, measured by flow cytometry and qPCR), the time to reach the highest concentration (Tmax) and the duration of cell survival in the patient;
3. PD index: proportion of peripheral blood plasma cells, concentration of free BCMA and cytokine release at each time point;
4. Quality of life assessment: the changes of subjects' quality of life before and after treatment were observed.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years old, gender is not limited;
2. Understand and know about this study and sign the informed consent voluntarily;
3. Patients diagnosed with recurrent/refractory plasma cell blood tumors must: a) have received at least 3 kinds of anti-plasma cell blood tumor therapy, including at least one proteasome inhibitor and one immunomodulator; b) documented progression within 12 months of treatment of the most recent antiplasmacytic blood tumor, or efficacy assessed as SD or PD within 60 days of treatment of the most recent antiplasmacytic blood tumor;
4. meet one of the following detection indicators: a) serum M protein ≥5g/L; b) Urine M protein ≥200mg/24h; c) Affected serum free light chain ≥100mg/L and abnormal serum free light chain ratio; d) Bone marrow plasma cell ratio ≥10%;
5. ECOG score is 0-2 points; 6, liver and kidney function, cardiopulmonary function meet the following requirements: a) blood creatinine ≤150umol/L, or creatinine clearance (estimated by Cockcroft Gaultra formula) ≥40ml/min (if the kidney function injury caused by rapid progression of the primary disease, the inclusion criteria can be appropriately relaxed, and the decision is made by the investigator); b) Total bilirubin ≤2×ULN; ALT≤3 x ULN, AST≤3 x ULN; c) Echocardiography showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥50%, and no serious arrhythmias; d) The subjects had no active pulmonary infection, and the blood oxygen saturation of indoor air was > 90%;

7. The subjects had no contraindications for peripheral blood monopexy, hemoglobin ≥60g/L, platelets ≥50×10^9/L, neutrophils ≥1×10^9/L; 8. Expected survival >12 weeks; 9. The urine pregnancy test of female subjects of childbearing age should be negative and not in the lactation period; Women or men of reproductive age were required to use effective contraception throughout the study.

Exclusion Criteria:

1. Have had severe rapid hypersensitivity to any of the drugs to be used in this study;
2. History of central nervous system (CNS) diseases, such as seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, neuropathy; Known active central nervous system (CNS) involvement or history of modification or clinical signs of multiple myeloma meningeal/spinal meningeal involvement;
3. Accompanied by other uncontrolled malignancies (except adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, and thyroid cancer after radical surgery);
4. The presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or any grade III (moderate) or grade IV (severe) heart disease (according to the New York Heart Society Functional Grading Method NYHA*); Patients with a history of myocardial infarction, angioplasty or stenting, unstable angina pectoris, or other clinically significant heart disease within 12 months prior to enrollment;
5. Previous patients with craniocerebral trauma, cerebrovascular accident, more serious cerebral ischemia or cerebral hemorrhage diseases;
6. The investigator determines that there are serious complications or diseases that increase the risk of the subject or affect the study, including but not limited to, for example, cirrhosis of the liver, recent major trauma, etc.;
7. Allogeneic hematopoietic stem cell transplantation performed within six months prior to screening, or hematopoietic stem cell transplantation performed during the screening period for any immunosuppressive treatment due to graft-versus-host disease;
8. Patients with autoimmune diseases, immune deficiencies or other immunosuppressants (other than low-dose glucocorticoids) are required;
9. Any uncontrolled active infection, including but not limited to active tuberculosis; Suspected uncontrollable fungal, bacterial, viral, or other infection prior to enrollment;
10. Received attenuated live vaccine within 4 weeks before anapheresis;
11. Subjects with active hepatitis (hepatitis B virus DNA >100IU/ml or hepatitis C virus RNA [HCVRNA] positive), syphilis, and other acquired and congenital immunodeficiency diseases, including but not limited to HIV-infected persons; People infected with CMV virus (CMV DNA test positive);
12. The subject has a history of alcoholism, drug abuse or mental illness;
13. Failure to follow the following treatment requirements needs to be excluded:

    A) Hormones: Subjects shall not receive more than 5mg of prednisone or other equivalent doses of corticosteroids and other immunosuppressive drugs within 72 hours prior to PBMC cell collection; B) Prior anti-tumor therapy (prior to PBMC monotherapy) : targeted therapy, epigenetic therapy or investigational drug therapy, or use of invasive investigational medical devices must have ended 14 days prior to PBMC cell collection or at least 5 half-lives (whichever is longer); Treatment of multiple myeloma with monoclonal antibodies ended at least 21 days before cell collection; Cytotoxic therapy should be completed at least 14 days before cell collection. Protease inhibitor treatment should end at least 14 days before cell collection. The immunomodulator should end at least 7 days before cell collection; C) Radiotherapy: must be completed no later than 4 weeks before PBMC cell collection, but if the radiotherapy field covered ≤ 5% of bone marrow reserve, participants were eligible to participate regardless of the radiotherapy end date; D) Anti-T cell antibody drugs (such as alenzumab) must be terminated 8 weeks before cell collection;
14. Researchers consider it inappropriate to participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To observe the number and incidence of adverse events after intravenous infusion of SENL103. | within 1 months after SENL103 infusion.
  The number, incidence and severity of all recorded adverse reactions, including cytokine release syndrome and neurotoxicity.

SECONDARY OUTCOMES:
Efficacy indicators | within 3 months after SENL103 infusion.
  To observe the efficacy of cell reperfusion, strict complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), disease stabilization (SD), disease-free progression-free survival (PFS rate), survival (OS) were adopted.
PD index | within 3 months after SENL103 infusion.
  the proportion of BCMA+ plasma cells in peripheral blood, the concentration of free BCMA and the release of cytokines at each time point;
PK index | within 3 months after SENL103 infusion.
  the highest concentration of SENL103 cells amplified in peripheral blood (Cmax, measured by flow cytometry and qPCR), the time to reach the highest concentration (Tmax) and the duration of cell survival in the patient;

CONTACTS AND LOCATIONS:
Overall Officials: Chunrui Li, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China